CLINICAL TRIAL: NCT07078656
Title: Effect of Video Training on Patients' Self-Efficacy After Colorectal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Gülçiçek Güngör, Graduate Student, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraYBU-SBF-GG-01
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Virtual reality video training; colorectal surgery; self-efficacy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Glasses (Experimental): Virtual reality glasses are a technological product that provides the human mind with the perception of real space and features of images arranged in a computer environment in 3 dimensions. It is also used as an educational tool, which is widely used in daily entertainment venues.
  Interventions: Behavioral: Postoperative management
- Control (No Intervention): In the control group, after obtaining permission with the "Informed Consent Form" one day before the surgery, the patients who agreed to participate in the study will fill out the "Patient Introduction Form" by the researchers, they will not receive any intervention and will be provided with routine nursing care provided in the hospital. The "Self-Efficacy Scale" will be applied when the patient comes for a check-up 10 days after discharge.

INTERVENTIONS:
Behavioral: Postoperative management — The patients who agreed to participate in the study will be asked to fill out a "Patient Introduction Form" by the researchers after obtaining permission from the experimental group with the "Informed Consent Form" the day before the surgery. On the 2nd day after laparoscopic colorectal surgery, virtual reality glasses will be worn by the patients and they will watch a 10-minute training video on the care of the patient after colorectal surgery. The training content will consist of topics such as dressing the surgical area, signs of infection in the surgical area (redness, swelling, discharge, color, temperature increase), pain management, unexpected situations (fever, nausea, abdominal pain, shivering, chan)
  Arms: Virtual Reality Glasses

SUMMARY:
The purpose of the study is to determine the effect of virtual reality video training on the self-efficacy of patients after colorectal surgery. Thus, correct planning can be provided for trainings that will provide information to patients according to their needs during the nursing care process.

Does virtual reality video training have an effect on participants' perceptions of self-efficacy after colorectal surgery? The researchers will conduct the self-efficacy survey on another group of participants without repeating the training to see the impact of the training.

Participants in the experimental group will receive training on the second postoperative day and they will apply a self-efficacy survey on the tenth day after discharge.

Participants in the control group will not receive training on the second postoperative day. They will complete a self-efficacy survey on the tenth day after discharge.

DETAILED DESCRIPTION:
The data obtained in the study will be evaluated in a computer environment using the IBM SPSS Version 22.0 package program. The conformity of the data to normal distribution will be assessed using the Kolmogorov-Smirnov test, and if the p value is p<0.05, Skewness and Kurtosis values will be examined. Descriptive statistics will be applied to sociodemographic variables. For intergroup comparisons of pre-test and post-test measurements of the experimental and control groups according to dependent variables, the significance test for the difference between two independent means will be used; for non-parametric data, the Mann Whitney U test will be used. For comparisons of pre-test and post-test measurements within the experimental and control groups according to dependent variables, the t-test for dependent groups will be used; for non-parametric data, the Wilcoxon test will be used. The results will be evaluated at a 95% confidence interval and a significance level of p<0.05.

ELIGIBILITY:
IInclusion Criteria:

* aged 18 and over
* aged 65 and under
* undergoing laparoscopic general surgery under general anesthesia
* with no vision, hearing, or perception problems
* with no communication problems
* without nausea, vomiting, dizziness, etc.
* with an ASA score of I, II, or III
* who voluntarily agreed to participate in the study

Exclusion Criteria:

* who have not undergone laparoscopic surgery
* who are hemodynamically unstable
* with an ASA score of IV
* with neurological or psychological problems
* Emergency and unplanned cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Self-Efficacy Scale in Colorectal Cancer Surgery | one week after registration up to 3 months
  This 16-question scale is scored using a Likert scale ranging from "not at all sure" to "very sure" (0-10). Questions include the ability to detect changes in the wound site (edema, redness, discharge, pain, discoloration, and increased temperature), timely medication use, dressing, seeking medical attention, regulating diet, detecting urinary changes, maintaining social relationships, and avoiding strenuous exercise. A higher score indicates an increase in self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Yılmazer, Ass. Prof., Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No